CLINICAL TRIAL: NCT06917664
Title: Treatment of Moderate Ischemic Mitral Regurgitation in Patients With Coronary Artery Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-I2M-C&T-B-070
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Ischemic Mitral Regurgitation; Angiotensin Receptor/Neprilysin Inhibitor
Keywords: coronary artery disease; ischemic mitral regurgitation; angiotensin receptor/neprilysin inhibitor
MeSH Terms: conditions — Coronary Artery Disease | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: isolated CABG (No Intervention)
- Sacubitril/valsartan therapy after isolated CABG (Experimental)
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril/valsartan therapy after isolated CABG
  Arms: Sacubitril/valsartan therapy after isolated CABG

SUMMARY:
This study aims to evaluate the effect of angiotensin receptor/neprilysin inhibitors (ARNI) on improving ischemic mitral regurgitation (IMR) in patients with coronary artery disease undergoing isolated coronary artery bypass grafting (CABG) through a randomized controlled clincial trial.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and voluntarily signed informed consent;
2. Received CABG and moderate IMR was diagnosed on two consecutive preoperative transthoracic echocardiography (according to 2021 ESC/EACTS Guidance Standards )

Exclusion Criteria:

1.Symptomatic hypotension and/or a SBP < 100 mmHg at screening; 2.Estimated GFR < 30 mL/min/1.73m2; 3.Serum potassium > 5 mmol/L at screening; 4.History of angioedema or unacceptable side effects while receiving ACE inhibitors or ARBs; 5.Patients receiving mitral valve intervention at the same time, or have participated in other clinical trials, or are unwilling to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
effective regurgitant orifice area (EROA) | 6 months postoperatively
  Change in EROA of mitral regurgitation evaluated by echocardiography from baseline to 6 months follow-up

SECONDARY OUTCOMES:
proportion of patients with moderate or higher IMR ,LVEF,LVESV,LVESVI,LVEDV,LVEDVI | 6 months postoperatively
  Proportion of patients with moderate or higher IMR; Left ventricular ejection fraction; Change of left ventricular end-systolic volume from baseline to 6 months follow-up; Change of left ventricular end-systolic volume index from baseline to 6 months follow-up; Change of left ventricular end-diastolic volume from baseline to 12 months follow-up; Change of left ventricular end-diastolic volume index from baseline to 12 months follow-up
major adverse cardiovascular and cerebrovascular events (MACCE) | 6 months postoperatively
  major adverse cardiovascular and cerebrovascular events (MACCE) defined as the composite of all-cause death, stroke, myocardial infarction, rehospitalization for heart failure, and repeat mitral valve surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Study Chair — China National Center for Cardiovascular Diseases
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tiemuerniyazi X, Chen L, He L, Yang Z, Huang S, Nan Y, Song Y, Yuan X, Hu Z, Zhao D, Zhao W, Feng W. The Role of Angiotensin Receptor/Neprilysin Inhibitor in Moderate Ischemic Mitral Regurgitation After Isolated Coronary Artery Bypass Grafting (ARNI-MIMIC): Study Protocol for a Randomized Controlled Trial. Am J Cardiol. 2025 Dec 1;256:102-106. doi: 10.1016/j.amjcard.2025.08.029. Epub 2025 Aug 21. PMID 40848924